CLINICAL TRIAL: NCT02125838
Title: Application of Endotracheal Intubation and Laryngeal Mask Supreme Without Neuromuscular Blocker in Laparoscopic Gynecologic Surgery
Brief Title: Laryngeal Mask Supreme During Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 859-GOA
Record Dates: First submitted 2014-01-31; First posted 2014-04-29 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Anaesthesia
Keywords: laryngeal mask Supreme; laparoscopic gynecologic surgery; Laryngeal mask during surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group ETT (Active Comparator): Group endotracheal tube In the endotracheal tube group for women no. 7-7.5 tube will use. ETT:Rüschelit, Teleflex Medical Sdn. Bhd. Malaysia. Ref:112482
  Interventions: Device: Endotracheal Tube
- Group LMS (Experimental): Laryngeal mask airway-supreme Group In the LMS group for <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) will insert.
  Interventions: Device: Laryngeal Mask Airway-Supreme

INTERVENTIONS:
Device: Laryngeal Mask Airway-Supreme — Group LM-S (Laryngeal Mask Airway-Supreme)Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.
  Other Names: Group LM-S
  Arms: Group LMS
Device: Endotracheal Tube — ETT
  Other Names: Group ETT
  Arms: Group ETT

SUMMARY:
Laryngeal mask (LM) use in gynecological laparoscopy, contrary to widespread opinion, does not increase the incidence of gastric aspiration, the failure of ventilation or the risk of pulmonary aspiration . LM is presented as an alternative to endo tracheal tube (ETT) in spontaneous or positive pressure ventilation (PPV) . LM has gained widespread popularity in England for gynecological laparoscopic procedures. In addition in many previous studies LM has been successfully shown to provide appropriate lung ventilation in laparoscopic surgical interventions .Miller et al. compared the use of ETT, LM-P laparoscopic gynecological interventions and identified advantages to LM use. The most important of these advantages was that, contrary to tracheal tube techniques for laparoscopic surgeries, use of supraglottic laryngeal devices or neuromuscular blocker agents (NBA) were not required during placement. Thus for laparoscopic surgeries, compared with the ETT technique, without the need for supraglottic laryngeal devices or muscular relaxants, it is easily placed and reduces the time spent in the operating room.

Our aim; to compare the use of LM-S and ETT without neuromuscular agents for laparoscopic gynecological intervention with positive pressure ventilation from a surgical viewpoint and in terms of effect on ventilation parameters.

Secondary aim, comparison of airway morbidity with endotracheal intubation and supraglottic.

DETAILED DESCRIPTION:
This prospective, randomized and double-blind study received permission from "Dokuz Eylül University Medical Faculty Non-Interventional Research Ethics Committee" and after obtaining patients' informed consent, 100 patients with American society of anesthesiologists (ASA) classification group I-II, between 18-65 years, undergoing elective laparoscopic gynecological surgery were included.

Patients were divided into:

Group 1=>ETT (50 patients) Group 2=>LM-S (50 patients) Patients and surgeons performing the operation were not aware of which airway device was used. The patients in the groups were determined by block randomized methods.

Patients taken to the surgical room were given standard monitoring (non-invasive blood pressure measurements, electrocardiogram, and peripheral oxygen saturation measurements) before anesthesia induction. For preoperative sedation 0.02 mg/kg midazolam IV was administered.

Patients were preoxygenated with 6 L/min oxygen for 3 minutes through a face mask.

For anesthesia induction after 2 minutes of 0.2 µg/kg/min remifentanil and 6 mg/kg/hr propofol infusion, IV 1-2 mg/kg propofol was administered. After induction patients were ventilated with 6 L/min 100% fraction of inspired oxygen inspired oxygen fraction oxygen through a face mask. Anesthesia depth was standardized in all patients using bispectral index monitoring. Bispectral index values were held between 40-60. Bispectral index values were maintained in this interval by increasing or decreasing propofol infusion by 1 mg/kg.

Airway devices were inserted by two researchers with more than 5 years experience.

During airway device placement according to patient reactions an extra dose of 0.5 mg/kg propofol was given if necessary.

Anesthetic maintenance was provided by 50% O2/air mixture with 0.1-0.4 µg/kg/min remifentanil and 50-150 µg/kg/hr (3-9 mg/kg/hr) propofol IV infusion.

Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.

After LM-S placement the cuff was inflated with air so as to have a pressure below 60 centimeters of water (cuff pressure manometer, Rusch, Germany). Two minutes after LM-S placement, before insufflation, 10 minutes after insufflation and trendelenburg position, before desufflation and before LM-S removal, cuff pressure was measured repeatedly and recorded. At the same time intervals in the ETT group, ETT cuff pressure was measured.

In the ETT group for women no. 7-7.5 tube was used. The ETT cuff was inflated until the leak sound ceased. It was measured with a manometer to remain between 20-30 centimeters of water.

Successful placement of LM or ETT was confirmed by square-shaped waves observed on the capnogram, easy ventilation of the respiration balloon and visible chest movements. After successful placement of the airway device, it was covered to prevent observation of which device was used.

The length of time for successful placement (duration from mouth opening to first successful ventilation), number of tries, and ease of placement were recorded. Ease of placement was evaluated by the anesthetist in charge of the airway as easy, hard or unsuccessful (alternative airway management).

In a situation where airway provision was unsuccessful after 3 tries, patients without placement of LM-S or who could not be intubated were switched to the other group and airway management was provided.

For oropharyngeal leak test after the expiratory valve was closed air was shut off, O2 was reduced to 3 L/min and the first pressure value when a leak sound was heard was recorded as the oropharyngeal leak pressure. To prevent exposure of the lungs to barotrauma, when the peak inspiratory pressure reached 40centimeters of water the expiratory valve was opened and the test was concluded. This test was repeated before peritoneal insufflation, 10 minutes later and immediately before desufflation and was completed by a researcher blind to the type of airway device inserted.

Positive pressure respiration was begun by using a ring system, 2-4 L/min fresh gas flow and 0.5 volume controlled 6-8 ml/kg tidal volume and 10 respirations/min frequency. Positive end expiratory pressure was not administered and I:E ratio was adjusted to 1:2. ETCO2 was held between 35-45 mmHg, if necessary first respiration frequency was increased then tidal volume was increased. Permission was given for CO2 insufflation for the laparoscopic intervention with peritoneal interior pressure of 15 mmHg.

Two minutes after LM-S or ETT placement, before insufflation, 10 minutes after insufflation and trendelenburg position, immediately before peritoneal desufflation and before airway device removal, ventilation parameters were evaluated.

Respiratory measurements to be recorded: Tidal volume (TV), respiration number (RN), peripheral oxygen saturation (SPO2), end-tidal carbon dioxide pressure (PETCO2), peak airway pressure (P peak), mean airway pressure (P mean) and expiration volume per minute (VE).

Hemodynamic measurements to be recorded: (simultaneous to the measurements above and additionally before induction) Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP) and heart rate (HR).

Evaluation related to gastric tube:

Immediately after airway device placement using either the LM-S drainage tube or in intubated patients using a 14 F orogastric probe within the airway, the stomach was reached and the gastric contents were aspirated. Ease of placement and amount of fluids aspirated were recorded. Ease of placement was classified by the person who inserted the orogastric probe as very easy, easy, difficult and very difficult.

The number of interventions with Verres needle, initial intra-abdominal pressure, duration to reach intra-abdominal pressure of 15 mmHg, and insufflated volume of CO2 were recorded. Sufficiency of pneumoperitoneum (sufficient/insufficient), and quality of airway provision were evaluated by the surgeon who was blind to the airway device used by giving points between 1-4.

Immediately after the intra-abdominal laparoscopic intervention and immediately before peritoneal insufflation was ended, gastric distension was evaluated by a surgeon blind to the airway device used between 0-10 (0=empty stomach, 10=distension obstructing the surgical field) and the difference between the scores at the start and end of the operation was recorded.

When the patient cooperated LM-S or ETT was removed and total anesthesia duration and peritoneal insufflation duration was recorded. Possible complications that could develop during airway device removal (coughing, vomiting, laryngeal stridor, laryngeal spasm or requirement for airway intervention) were recorded.

After laryngeal supra glottic airway device removal the presence of blood was evaluated as

1. no blood
2. trace amounts of blood
3. clear amount of blood Revived patients were taken to the recovery unit and a blind researcher evaluated the patients' throat pain, hoarseness and presence of difficulty swallowing in the 1st and 24th hours. To evaluate throat pain the visual analogue scale was used.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification group I-II
* Between 18-65 years
* Undergoing elective laparoscopic gynecological surgery

Exclusion Criteria:

* Individuals with any neck and upper respiratory pathology
* Individuals at risk of gastric content regurgitation/aspiration (previous upper gastrointestinal surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcer, full stomach, pregnancy)
* Individuals with low pulmonary compliance or high airway resistance (chronic lung diseases)
* Obese patients (BMI >35)
* Individuals with sore throat, dysphagia and dysphonia
* Individuals with possibility or history of difficult airway
* Operation time planned for more than 4 hours

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SULE OZBİLİGİN, M.D., Principal Investigator — STUDY DESİGN
Locations (1):
- Sule Ozbilgin, Izmi̇r, Narlıdere, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group ETT: Group ETT (Endotracheal tube Group). In the ETT group for women no. 7-7.5 tube will use. ETT:Rüschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
  Endotracheal Tube: ETT
- Group LMS: Group LM-S (Laryngeal mask supreme Group) For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) will insert.
  Laryngeal Mask Airway-Supreme: Group LM-S (laryngeal mask group)Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.
Period: Overall Study
Arm/Group | Group ETT | Group LMS
Started | 54 (Lost to follow-up (n= 4 ) Turned to laparotomy (Adhesions)(n= 2) NBA used (n= 2)) | 54 (Lost to follow-up (n= 4 ) Turned to laparotomy (Adhesions) (n= 2) NBA used (n= 2))
Completed | 50 (Analysed (n=50 )) | 50 (Analysed (n=50 ))
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group ETT | Group LMS | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 54 | 108
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Asses to Ventilation Parameters
Description: tidal volume (ml) at certain time intervals T1= 2 minutes after airway device insertion T2= 10 minutes after insufflation T3= Before desufflation T4= Before removal of airway device
Time Frame: intraoperative period
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
ml
  T1 | 451.8 (62.6) | 437.1 (62.0)
  T2 | 457.2 (57.1) | 443.6 (61.5)
  T3 | 462 (63.0) | 451.3 (58.5)
  T4 | 464.8 (58.7) | 448.1 (53.9)

2. Secondary Outcome: Quality of View According to Surgeon by Rate Scale
Description: Quality of surgical view will be assessed with points from 1 to 4 by the surgeon blind to the airway device by Rate Scale.
  Grade of quality of view were evaluated between 1-4 points (1-poor to 4-excellent)
Time Frame: intraoperative period
Measure: Number; unit: percentage of participants
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
percentage of participants
  Grade I | 0 | 0
  Grade II | 4 | 2
  Grade III | 20 | 22
  Grade IV | 76 | 76

3. Secondary Outcome: Evaluation of Gastric Distention
Description: To provide the adequate gastric distention of either the LM-Supreme or the tracheal tube, as assigned. Gastric distension was evaluated by a surgeon blind to the airway device used between 0-10 (0=empty stomach, 10=distension obstructing the surgical field)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
units on a scale | 2.98 (2.37) | 3.144 (1.98)

4. Secondary Outcome: Ease of Orogastric Tube Placement Classification
Description: Ease of placement was classified by the person who inserted the orogastric tube as very easy, easy, difficult or very difficult.
Time Frame: Baseline
Population: Ease of placement was classified by the person who inserted the orogastric tube as very easy, easy, difficult or very difficult.
Measure: Number; unit: participants
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
participants
  very easy | 19 | 38
  easy | 23 | 10
  diffucult | 7 | 2
  very diffucult | 1 | 0

5. Secondary Outcome: Haemodynamic Response to Insertion of Airway Device
Description: Systolic blood pressure and heart rate at two minutes after LM-S placement, before insufflation, 10 minutes after insufflation and trendelenburg position, before desufflation and before LM-S removal .
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Post-operative Sore Throat
Description: Patients were asked about the presence of sore throat - defined as the presence of constant pain in the throat, independent of swallowing, 1 hr and 24 hr after the end of surgery.
Time Frame: Baseline
Reporting Status: Not Posted

7. Primary Outcome: Asses to Peak Pressure
Description: peak pressure (cmH20) at certain time intervals T1= 2 minutes after airway device insertion T2= 10 minutes after insufflation T3= Before desufflation T4= Before removal of airway device
Time Frame: intraoperative period
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
cmH20
  T1 | 13.1 (3.5) | 11.8 (2.9)
  T2 | 19.5 (4.7) | 18.5 (4.5)
  T3 | 18.7 (5.6) | 17.5 (4.4)
  T4 | 14.8 (3.2) | 13.4 (3.4)

8. Primary Outcome: Asses to Mean Pressure
Description: mean pressures within the times below (cmH20) T1= 2 minutes after airway device insertion T2= 10 minutes after insufflation T3= Before desufflation T4= Before removal of airway device
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Group ETT | Group LMS
Number analyzed (Participants) | 50 | 50
cmH20
  T1 | 6.2 (1.7) | 5.9 (1.5)
  T2 | 8.5 (2.1) | 8.1 (3.1)
  T3 | 8.0 (1.8) | 7.5 (1.5)
  T4 | 6.6 (1.3) | 6.1 (1.1)

ADVERSE EVENTS:
Arm/Group | Group ETT | Group LMS
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No